# *ICF*

### Incapacitated subjects

## **MOSART-study**

Neurotoxic adverse effects of morphine and oxycodone in continuous subcutaneous infusion for treatment of pain in terminal patients with diminished renal function: a Randomized Controlled Trial.

Version number: 2, date 2017.08.18

# Informatie voor de vertegenwoordiger voor deelname aan medisch-wetenschappelijk onderzoek

### **MOSART-studie**

Een onderzoek naar verschillen in bijwerkingen tussen morfine en oxycodon bij continue toediening voor behandeling van pijn bij personen in de stervensfase.

Officiële titel: Neurotoxische bijwerkingen van morfine en oxycodon voor continue subcutane infusie ter behandeling van pijn bij terminale patiënten met een verminderde nierfunctie: een Randomized Controlled Trial.

### Inleiding

Geachte heer/mevrouw,

U vertegenwoordigt een persoon die zelf niet meer in staat is om beslissingen te nemen. Wij benaderen u met de vraag voor deelname van degene die u vertegenwoordigt aan een medisch-wetenschappelijk onderzoek. Meedoen is vrijwillig. Om mee te doen is wel uw schriftelijke toestemming nodig.

U ontvangt deze brief omdat de behandelend arts van persoon die u vertegenwoordigt heeft vastgesteld dat continue toediening van een opioïd (een sterke pijnstiller) nodig is om pijn in de laatste levensfase te behandelen.

Voordat u beslist of hij/zij meedoet aan dit onderzoek, krijgt u uitleg over wat het onderzoek inhoudt. Lees deze informatie rustig door en vraag de onderzoeker om uitleg als u vragen heeft. U kunt ook de onafhankelijke deskundige, die aan het eind van deze brief genoemd wordt, om aanvullende informatie vragen. En u kunt er ook over praten met uw partner, vrienden of familie.

Verdere informatie over meedoen aan zo'n onderzoek staat in de bijgevoegde brochure 'Medisch-wetenschappelijk onderzoek'.

### 1. Algemene informatie

Dit onderzoek is opgezet door het Expertisecentrum Palliatieve Zorg van het Maastricht Universitair Medisch Centrum en wordt gedaan door artsen en onderzoekers in verschillende verpleeghuizen en hospices. Voor dit onderzoek zijn in totaal 234 proefpersonen nodig.

Dit onderzoek wordt mede mogelijk gemaakt door een subsidie van ZonMw en cofinanciering door Envida en het Maastricht Universitair Medisch Centrum.

De medisch ethische toetsingscommissie van het azM/UM (METC azM/UM) heeft dit onderzoek goedgekeurd. Algemene informatie over de toetsing van onderzoek vindt u in de brochure 'Medisch-wetenschappelijk onderzoek'.

### 2. Doel van het onderzoek

Het doel van dit onderzoek is het vergelijken van bepaalde bijwerkingen bij het continu toedienen van morfine of oxycodon voor pijnbestrijding bij patiënten in de laatste levensfase met een verminderde nierfunctie.

### 3. Achtergrond van het onderzoek

In de laatste levensfase komt pijn vaak voor. De 'morfine-pomp' is een veel gebruikte behandeling voor deze pijn. Hierbij wordt continu een hoeveelheid morfine toegediend via een klein onderhuids naaldje (dit noemen we subcutane infusie). Een andere mogelijkheid is dat om de vier uur een vergelijkbare hoeveelheid morfine via dit onderhuidse naaldje wordt toegediend. Beide methodes werken even goed.

Het is echter de vraag of morfine wel het meest geschikte middel is in deze situatie. Door achteruitgang van lichaamsfuncties in deze laatste levensfase, waaronder vermindering van de nierfunctie, kunnen afbraakproducten van morfine zich namelijk gaan opstapelen in het lichaam. We vermoeden dat door deze opstapeling van afbraakproducten mogelijk bijwerkingen zouden kunnen ontstaan, zoals onrust en/of verwardheid (in medische termen wordt dit een delier genoemd) of zelfs toegenomen pijnbeleving. Dit zou dan kunnen leiden tot een sterfbed met toenemende onrust en/of pijn, terwijl we juist het tegenovergestelde proberen te bereiken.

Oxycodon is een middel dat vergelijkbaar is met morfine. Het zijn beide sterke pijnstillers, die we opioïden noemen. Oxycodon wordt net als morfine al langdurig in de praktijk toegepast en heeft geen nadelen ten opzichte van morfine. De keuze voor één van beide middelen berust in de praktijk vaak op de persoonlijke voorkeur van de arts. Oxycodon heeft echter minder opstapelende afbraakproducten dan morfine. We denken dat hierdoor in theorie bij oxycodon minder van de genoemde vervelende bijwerkingen zouden kunnen optreden.

Dat is echter op dit moment alleen nog maar een theorie, die nog nooit eerder goed is onderzocht. Het is hierdoor nog onbekend of oxycodon in de praktijk ook echt minder van de genoemde bijwerkingen geeft dan morfine. Dat willen we met dit onderzoek gaan vergelijken. Met de uitkomsten van dit onderzoek zouden we een belangrijke bijdrage kunnen leveren aan het verbeteren van de kwaliteit van zorg voor mensen in de laatste levensfase.

### 4. Wat meedoen inhoudt

Deelname aan het onderzoek duurt net zo lang als de behandeld arts nodig vindt dat de pijnstiller toegediend krijgt. In de praktijk is dit vrijwel altijd tot aan het overlijden.

### Geschiktheidsonderzoek

Om deel te kunnen nemen aan dit onderzoek hebben wij uiteraard toestemming nodig. De persoon die u vertegenwoordigd, is echter niet meer in staat om zelf beslissingen te nemen. Daarom vragen wij u, als vertegenwoordiger van deze persoon, om toestemming voor deelname aan het onderzoek. Hiervoor dient het toestemmingsformulier door u ondertekent te worden. Als u uw toestemming heeft gegeven, zullen we vervolgens eerst bepalen of degen die u vertegenwoordigt ook daadwerkelijk geschikt is om mee te doen. Hiervoor hebben we zijn/haar medische gegevens nodig van de behandelend arts. Daarnaast zullen we bij het eerste bezoek eenmalig bloed moeten prikken. Dat is nodig om de nierfunctie te bepalen. Als uit het bloedonderzoek blijkt dat de nierfunctie niet verminderd is, stopt op dat moment de verdere deelname aan het onderzoek.

Als u dit niet wilt, kan de persoon die u vertegenwoordigt niet meedoen aan dit onderzoek.

### Behandeling

De ene helft van de studiedeelnemers krijgt morfine, de andere helft oxycodon. Loting bepaalt welke van deze twee pijnstillers degene die u vertegenwoordigt krijgt. Dit middel zal na de loting gewoon door zijn/haar eigen arts worden voorgeschreven. Hij/zij blijft verder ook volledig de normale zorg van zijn/haar eigen arts ontvangen, zoals hij/zij dat anders ook zou krijgen.

De onderzoeksverpleegkundige die gedurende het onderzoek steeds bij hem/haar langs komt, weet niet in welke groep hij/zij zit. Zo wordt de onderzoeksverpleegkundige niet beïnvloed bij het uitvoeren van de metingen. Het is dan ook belangrijk dat u hem/haar niet vertelt welke van de twee pijnstillers de persoon die u vertegenwoordigt krijgt.

Algemene informatie hierover vindt u in de brochure 'Medisch-wetenschappelijk onderzoek'.

### Bezoeken en metingen

Wij komen de persoon die u vertegenwoordigd bezoeken in zijn/haar eigen kamer in het verpleeghuis of hospice waar hij/zij verblijft. Hij/zij hoeft dus zelf niet te reizen. Deze bezoeken worden uitgevoerd door (één van) onze onderzoeksverpleegkundigen.

Bij het eerste bezoek zal de onderzoeksverpleegkundige eenmalig één buisjes bloed afnemen. Dit is om de nierfunctie te bepalen.

Vervolgens zal de onderzoeksverpleegkundige drie keer per week een bezoek brengen. Een bezoek duurt ongeveer tien minuten. Er zal dan het volgende gebeuren:

- Wij vragen degene die u vertegenwoordigd om aan te geven hoeveel pijn hij/zij heeft. Als hij/zij niet (meer) in staat is om dit aan te geven, kijken wij of we kenmerken van pijn bij hem/haar kunnen zien.
- Wij strijken kort met een watje over de onderarmen en vragen of dit pijnlijk aanvoelt. Als hij/zij niet (meer) in staat is om dit aan te geven, kijken wij of we hem/haar kenmerken van een pijnlijke reactie kunnen zien.
- Wij laten kort een scherpe naald op de onderarmen rusten (zonder hem/haar te prikken uiteraard) en vragen of dit pijnlijk aanvoelde. Als hij/zij niet (meer) in staat is om dit aan te geven, kijken wij of we kenmerken van een pijnlijke reactie bij hem/haar kunnen zien.

Daarnaast zal de onderzoeksverpleegkundige bij elk bezoek de volgende informatie verzamelen bij het verzorgend personeel van de afdeling:

- De medicatie die op dat moment gebruikt wordt.
- Of zij tekenen van een delier (onrust/verwardheid) hebben waargenomen.
- Of zij nog andere bijwerkingen hebben waargenomen.

Na het overlijden zouden wij graag een naaste van degene die u vertegenwoordigd, die veel bij hem/haar aanwezig was in de periode rond het overlijden, telefonisch willen benaderen voor een interview door de onderzoeker over hoe deze persoon deze periode heeft ervaren. Als vertegenwoordiger kunt u dit zelf zijn, maar dit mag ook een andere persoon zijn. Dit telefonisch interview mag alleen plaatsvinden als zowel u, als de desbetreffende naaste hier toestemming voor geven.

### 5. Wat wordt er van de persoon die u vertegenwoordigt verwacht

Om het onderzoek goed te doen verlopen, is het belangrijk dat hij/zij zich aan de volgende afspraken houdt.

De afspraken zijn dat hij/zij:

- het onderzoeksmiddel toe laat dienen volgens het voorschrift van uw arts.
- niet ook nog aan een ander medisch-wetenschappelijk onderzoek meedoet.
- afspraken voor bezoeken die worden gaan worden, respecteert.
- de onderzoeksverpleegkundige(n) niet vertelt welke van de twee pijnstillers degene die u vertegenwoordigt krijgt.

### 6. Mogelijke bijwerkingen

De onderzoeksmiddelen morfine en oxycodon kunnen bijwerkingen geven.

Deze bijwerkingen komen vaak voor (bij 1 op de 10 mensen of meer):

- Obstipatie. De behandelend arts kan hiervoor een laxeermiddel voorschrijven.
- Misselijkheid en braken. Dit verdwijnt meestal na een paar dagen. De behandelend arts kan tijdelijk een middel tegen de misselijkheid voorschrijven.
- Slaperigheid of sufheid. Dit verdwijnt meestal na een paar dagen.
- Droge mond. De behandelend arts kan middelen voorschrijven die deze klachten kunnen verminderen.

Deze bijwerkingen komen voor, maar niet zo vaak:

- Jeuk. De behandelend arts kan een middel voorschrijven dat deze klachten kan verminderen.
- Onvolledige blaaslediging (blaasretentie). Een blaaskatheter kan de klachten hiervan wegnemen.

De onderzoeksmiddelen kunnen ook bijwerkingen hebben die nog onbekend zijn.

Meer informatie over oxycodon en morfine staat in de bijsluiters. Doet u mee aan het onderzoek? Dan kunt u uw behandelend arts hierom vragen.

### Metingen

Een bloedafname kan pijn doen of een bloeduitstorting geven.

Het strijken met een watje over de huid of het plaatsen van een scherpe naald op de huid kan mogelijk kortdurend een pijnlijke reactie oproepen bij het uitvoeren hiervan.

### 7. Mogelijke voor- en nadelen

Het is belangrijk dat u de mogelijke voor- en nadelen goed afweegt voordat u besluit dat de persoon die u vertegenwoordigt mee doet.

### Voordelen

Wanneer hij/zij door loting in de morfine-groep wordt ingedeeld, heeft hij/zij zelf geen voordeel van meedoen aan dit onderzoek. Zijn/haar deelname kan wel bijdragen aan meer kennis over de behandeling van pijn in de terminale fase.

Wanneer hij/zij door loting in de oxycodon-groep wordt ingedeeld, kan de kans kleiner worden dat bij hem/haar onrust/verwardheid (een delier) of een toegenomen pijnbeleving optreedt, maar zeker is dat niet.

### Nadelen

Een nadeel van meedoen aan het onderzoek kan zijn dat hij/zij mogelijk ongemakken ondervindt van de metingen in het onderzoek.

Deelname aan het onderzoek betekent ook:

- dat hij/zij in zijn/haar laatste levensperiode drie maal per week bezoek krijgt van een 'vreemde' onderzoeksverpleegkundige;
- dat hij/zij tijdens dit bezoek 5 tot 10 minuten van zijn tijd kwijt is;
- dat hij/zij afspraken heeft waaraan hij/zij zich moet houden.

Al deze zaken zijn hiervoor onder punt 4, 5 en 6 beschreven. Uiteraard zullen wij ons maximaal inspannen om de overlast voor u tot een minimum te beperken.

### 8. Verzet van degene die u vertegenwoordigt

Het kan zijn dat degene die u vertegenwoordigt zich tijdens het onderzoek verzet (niet meewerkt). De onderzoeker moet het onderzoek dan direct stoppen. Het is moeilijk om precies te omschrijven wat verzet is. Voor de start van het onderzoek wordt met u overlegd wat als verzet wordt gezien.

De onderzoeker zal zich houden aan de Gedragscode verzet geriatrische patiënten.

# 9. Als u niet wilt dat degene die u vertegenwoordigt meedoet of als u wilt dat er gestopt wordt met het onderzoek

U beslist zelf of de persoon die u vertegenwoordigt meedoet aan het onderzoek. Deelname is vrijwillig.

Als u niet wilt dat hij/zij meedoet, wordt hij/zij op de gebruikelijke manier behandeld voor de pijn. Het feit dat hij/zij voor deelname aan dit onderzoek in aanmerking komt, betekent dat zijn/haar behandelend arts al heeft vastgesteld dat deze behandeling het beste kan plaatsvinden met continue toediening van een opioïd. De behandelend arts bepaalt dan zelf welk opioïd hij/zij toegediend krijgt.

Als u besluit dat hij/zij wel meedoet, kunt u zich altijd bedenken en deelname toch stoppen, ook tijdens het onderzoek. Hij/zij wordt dan weer op de gebruikelijke manier behandeld voor de pijn. U hoeft niet te zeggen waarom u wilt dat er gestopt. Wel moet u dit direct melden aan de onderzoeker.

De gegevens die tot dat moment zijn verzameld, worden gebruikt voor het onderzoek.

Als er nieuwe informatie over het onderzoek is die belangrijk voor u is, laat de onderzoeker dit aan u weten. U wordt dan gevraagd of u wilt dat de persoon die u vertegenwoordigt blijft meedoen.

### 10. Einde van het onderzoek

De deelname aan het onderzoek stopt als

- uit het bloedonderzoek blijkt dat de nierfunctie niet verminderd is;
- alle bezoeken zoals beschreven onder punt 4 voorbij zijn;
- · u zelf kiest dat er gestopt wordt;
- de behandelend arts het niet langer nodig vindt dat er met een opioïd behandeld wordt;
- de onderzoeker het beter vindt voor de persoon die u vertegenwoordigt om te stoppen;
- de behandelend arts het beter vindt voor de persoon die u vertegenwoordigt om te stoppen;
- de persoon die u vertegenwoordigt verhuist buiten de deelnemende instellingen;
- het Expertisecentrum Palliatieve Zorg MUMC+, ZonMw, Envida, de overheid of de beoordelende medisch ethische toetsingscommissie besluiten om het onderzoek te stoppen.

Het hele onderzoek is afgelopen als alle deelnemers zijn overleden of om de overige genoemde redenen met deelname aan het onderzoek zijn gestopt.

Morfine en oxycodon zijn gangbare middelen, die door uw eigen behandelend arts worden voorgeschreven. Wanneer u besluit dat u wilt dat degene die u vertegenwoordigd stopt met deelname aan het onderzoek, blijft hierdoor de medicatie die u gebruikt heeft tijdens het onderzoek naderhand beschikbaar via uw behandelend arts. Uiteraard alleen wanneer de behandelend arts het gebruik van deze middelen voor deze persoon nodig acht. De onderzoeker zal met u praten over de mogelijkheden voor verdere medische zorg.

### 11. Gebruik en bewaren van gegevens en lichaamsmateriaal

Voor dit onderzoek is het nodig dat bloed en medische en persoonsgegevens worden verzameld en gebruikt. Elke proefpersoon krijgt een code die op het bloedbuisje en de gegevens komt te staan. De naam en andere persoonsgegevens worden weggelaten.

### De gegevens van de persoon die u vertegenwoordigt

Alle gegevens blijven vertrouwelijk. Alleen de onderzoekers en de onderzoeksverpleegkundigen weten welke code de persoon die u vertegenwoordigt heeft. De sleutel voor de code blijft bij de onderzoeker. Ook in rapporten over het onderzoek wordt alleen die code gebruikt.

Sommige mensen mogen de medische en persoonsgegevens inzien. Dit is om te controleren of het onderzoek goed en betrouwbaar uitgevoerd is. Algemene informatie hierover vindt u in de brochure 'Medisch-wetenschappelijk onderzoek'.

Mensen die de gegevens kunnen inzien zijn: het onderzoeksteam, een controleur die door de uitvoerder van het onderzoek is ingehuurd en de Inspectie voor de Gezondheidszorg. Zij

houden de gegevens geheim. Als u de toestemmingsverklaring ondertekent, geeft u toestemming voor het verzamelen, bewaren en inzien van de medische en persoonsgegevens van de persoon die u vertegenwoordigt.

De onderzoeker bewaart deze gegevens 15 jaar.

### Lichaamsmateriaal van de persoon die u vertegenwoordigt

Het bloed dat afgenomen is, wordt door de onderzoeksverpleegkundige naar het Centraal Diagnostisch Laboratorium van het MUMC+ gebracht. Daar wordt het enkel gebruikt voor het bepalen van uw nierfunctie. Na deze bepaling wordt het bloed niet bewaard of voor andere doeleinden gebruikt.

Algemene informatie over de registratie van onderzoeken vindt u in de brochure 'Medischwetenschappelijk onderzoek'

### 12. Verzekering voor proefpersonen

Voor iedereen die meedoet aan dit onderzoek is een verzekering afgesloten. De verzekering dekt schade door het onderzoek. Niet alle schade is gedekt. In bijlage B vindt u meer informatie over de verzekering. Daar staat ook aan wie u schade kunt melden.

### 13. Informeren behandelend arts en apotheker

Wij sturen de behandelend arts en apotheker van het verpleeghuis of hospice waar degene die u vertegenwoordigt verblijft altijd een brief om te laten weten dat hij/zij meedoet aan het onderzoek. Dit is voor zijn/haar eigen veiligheid. Als u dit niet goed vindt, kan hij/zij niet meedoen aan dit onderzoek.

### 14. Geen vergoeding voor meedoen

Deelname aan dit onderzoek kost u en de persoon die u vertegenwoordigt niets. U of degene die u vertegenwoordigt worden niet betaald voor het meedoen aan dit onderzoek.

### 15. Heeft u vragen?

Bij vragen kunt u contact opnemen met de onderzoeker. Voor onafhankelijk advies over meedoen aan dit onderzoek kunt u terecht bij de onafhankelijke arts. Hij weet veel over het onderzoek, maar heeft niets te maken met dit onderzoek.

Bij klachten kunt u het beste terecht bij de klachtencommissie van uw instelling. Alle gegevens vindt u in **bijlage A**: Contactgegevens.

### 16. Ondertekening toestemmingsformulier

Wanneer u voldoende bedenktijd heeft gehad, wordt u gevraagd te beslissen over deelname van de persoon die u vertegenwoordigt aan dit onderzoek. Indien u toestemming geeft, zullen wij u vragen dit op de bijbehorende toestemmingsverklaring schriftelijk te bevestigen. Door uw schriftelijke toestemming geeft u aan dat u de informatie heeft begrepen en instemt met deelname van de persoon die u vertegenwoordigt aan het onderzoek.

Het handtekeningenblad overhandigt u aan de behandelend arts. Dit zal vervolgens door de onderzoeker opgehaald en bewaard worden. U krijgt een kopie of een tweede exemplaar van deze toestemmingsverklaring.

Indien u toestemming heeft gegeven dat een naaste na het overlijden van degene die u vertegenwoordigd, benaderd mag worden voor een telefonisch interview, zal ook aan deze persoon gevraagd worden om een toestemmingsverklaring hiervoor te ondertekenen. Ook deze toestemmingsverklaring kan overhandigd worden aan de behandelend arts en zal vervolgens door de onderzoeker opgehaald en bewaard worden.

Dank voor uw aandacht.

### Bijlagen bij deze informatie

- A. Contactgegevens voor Envida
- B. Informatie proefpersonenverzekering
- C. Toestemmingsformulier proefpersoon
- D. Toestemmingsformulier nabestaande
- E. Brochure 'Medisch-wetenschappelijk onderzoek. Algemene informatie voor de proefpersoon' (versie mrt 2017)

### Bijlage A: contactgegevens voor Envida

Onderzoeker: Drs. M.J.M. (Mark) Martens

specialist ouderengeneeskunde, Envida

consulent palliatieve zorg, Expertisecentrum Palliatieve Zorg MUMC+

Tel.: 043 - 85093084

Onafhankelijk arts: Dr. med. M.N. (Markus) Janssen, FIPP

anesthesioloog/pijngeneeskundige MUMC+

Tel.: 043 - 3875606

Klachten: Elly Wijnen

klachtenfunctionaris Stichting Envida Tel.: 0900 - 2233440 / 06 – 23863129

E-mail: klachten@envida.nl

### Bijlage B: INFORMATIE PROEFPERSONENVERZEKERING

#### **VERZEKERINGSVERKLARING**

voor het hierna te noemen wetenschappelijk onderzoek

Titel: Neurotoxic adverse effects of morphine and oxycodone in continuous subcutaneous infusion for treatment of pain in terminal patients with diminished renal function: a Randomized Controlled Trial.

Voor iedereen die meedoet aan dit onderzoek, heeft het academisch ziekenhuis Maastricht, hierna te noemen azM, een verzekering afgesloten. De verzekering dekt schade door deelname aan het onderzoek. Dit geldt voor schade tijdens het onderzoek of binnen vier jaar na het einde ervan. Schade moet u binnen die vier jaar aan de verzekeraar hebben gemeld.

De verzekering dekt niet alle schade. Onderaan deze tekst staat in het kort welke schade niet wordt gedekt. Deze bepalingen staan in het Besluit verplichte verzekering bij medisch-wetenschappelijk onderzoek met mensen. Dit besluit staat op www.ccmo.nl, de website van de Centrale Commissie Mensgebonden Onderzoek (zie 'Bibliotheek' en dan 'Weten regelgeving').

Bij schade kunt u direct contact leggen met de verzekeraar:

De verzekeraar van het onderzoek is:

Naam: CNA Insurance Company Ltd.

Adres: World Trade Centre, Strawinskylaan 703, 1077 XX Amsterdam

Telefoonnummer: 020-5737272

Polisnummer: 10174880

Contactpersoon: Esther van Herk, Snr Claims Examiner

E-mail: Esther.VanHerk@cnaeurope.com

Telefoonnummer: 020-5737274

De verzekering biedt een dekking van ten minste € 650.000 per proefpersoon en ten minste € 5.000.000 voor het hele onderzoek (en ten minste € 7.500.000 per jaar voor alle onderzoeken van het azM).

De verzekering dekt de volgende schade niet:

- schade door een risico waarover u in de schriftelijke informatie bent ingelicht. Dit geldt niet als het risico zich ernstiger voordoet dan was voorzien of als het risico heel onwaarschijnlijk was;
- schade aan uw gezondheid die ook zou zijn ontstaan als u niet aan het onderzoek had meegedaan;
- schade door het niet (volledig) opvolgen van aanwijzingen of instructies;
- schade aan uw nakomelingen, als gevolg van een negatief effect van het onderzoek op u of uw nakomelingen;
- schade door een bestaande behandelmethode bij onderzoek naar bestaande behandelmethoden.

### Bijlage C: Toestemmingsformulier vertegenwoordiger

| МО | SART-stu | die | |
|---|---|---|---|
| | | gd om toestemming te geven voor<br>nschappelijke onderzoek: | deelname van de volgende persoon aan dit |
| Naa | am proefpe | ersoon: | Geboortedatum:// |
| - | Mijn vrag | · · | voordiger gelezen. Ook kon ik vragen stellen.<br>had genoeg tijd om te beslissen of deze |
| - | | at meedoen vrijwillig is. Ook weet<br>soon toch niet meedoet. Daarvoor | ik dat ik op ieder moment kan beslissen dat hoef ik geen reden te geven. |
| - | _ | eeghuis of hospice waar deze pers | an de behandelend arts en de apotheker van soon verblijft, dat deze persoon meedoet aan |
| - | verpleegl | , , | n informatie bij de behandelend arts in het<br>n verblijft over de medische voorgeschiedenis,<br>bruik van deze persoon. |
| - | | at sommige mensen de gegevens<br>staan vermeld in deze informatieb | van deze persoon kunnen inzien. Die rief. |
| - | persoon | | de gegevens en het bloedmonster van deze<br>ie in de informatiebrief (zie ook sectie 4 onder |
| - | _ | estemming om de gegevens op dek te bewaren. | e onderzoek-locatie nog 15 jaar na dit |
| - | • | iken voor controle of verdere anal | derzoek oplevert eventueel in de toekomst te<br>yse in het kader van wetenschappelijk |
| - | lk geef | □ wel<br>□ niet | |
| | | , | den van deze persoon telefonisch benaderd te<br>de onderzoeker over hoe ik de periode rond |
| | | recht voor om af te zien van dit | n heb ervaren. Ik behoud me te allen tijde het interview zonder opgave van reden. |

- Ik ga ermee akkoord dat deze persoon meedoet aan dit onderzoek.

| Naam wettelijk vertegenwoordiger: | |
|---|---|
| Relatie tot de proefpersoon: | |
| Handtekening: | Datum: / / |
| Ik verklaar hierbij dat ik deze persoon/personen volledig heb ge<br>genoemde onderzoek. | eïnformeerd over het |
| Als er tijdens het onderzoek informatie bekend wordt die de toe<br>vertegenwoordiger zou kunnen beïnvloeden, dan breng ik hem<br>hoogte. | - |
| Naam onderzoeker (of diens vertegenwoordiger):<br>Handtekening: | Datum: / / |
| <indien toepassing="" van=""> Aanvullende informatie is gegeven door (indien van toepassing</indien> | |
| Naam: | <i>)</i> . |
| Functie:<br>Handtekening: | Datum: / / |
| * Doorhalen wat niet van toepassing is. | |

De proefpersoon krijgt een volledige informatiebrief mee, samen met een kopie van het getekende toestemmingsformulier.

Proefpersoneninformatie

### Bijlage D: toestemmingsformulier nabestaande

#### **MOSART-studie**

Een naaste van u neemt deel aan de MOSART-studie. Hij/zij heeft aangegeven toestemming te geven om na zijn/haar overlijden u te mogen benaderen voor een telefonisch interview door de onderzoeker over hoe u deze periode rond het overlijden ervaren hebt. Uiteraard benaderen wij u alleen hiervoor indien ook u hiervoor toestemming geeft.

- Ik heb de informatiebrief gelezen. Ook kon ik vragen stellen. Mijn vragen zijn voldoende beantwoord. Ik had genoeg tijd om te beslissen of ik meedoe.
- Ik weet dat meedoen vrijwillig is. Ook weet ik dat ik op ieder moment kan beslissen om toch niet mee te doen of te stoppen met het interview. Daarvoor hoef ik geen reden te geven.
- Ik weet dat sommige mensen mijn gegevens kunnen inzien. Die mensen staan vermeld in deze informatiebrief.
- Ik geef toestemming voor het verzamelen en gebruiken van mijn gegevens op de manier en voor de doelen die in de informatiebrief staan (zie ook sectie 4).
- Ik geef toestemming om mijn gegevens op de onderzoek-locatie nog 15 jaar na dit onderzoek te bewaren.
- Ik geef toestemming om de data die dit onderzoek oplevert eventueel in de toekomst te hergebruiken voor controle of verdere analyse in het kader van wetenschappelijk onderzoek.
- Ik wil meedoen aan dit interview.

| Naam nabestaande: | |
|-------------------|-------------|
| Handtekening: | Datum : / / |

| Proefpersoneninformatie | |
|---|---|
| lk verklaar dat ik deze proefpersoon volledig heb geïnformeerd over het genoemde onderzoek. | |
| Als er tijdens het onderzoek informatie bekend wordt die de toestemming van de proefpersoon zou kunnen beïnvloeden, dan breng ik hem/haar daarvan tijdig op de hoogte. | |
| Naam onderzoeker (of diens vertegenwoordiger): | |
| Handtekening: | Datum: / / |
| <pre><indien toepassing="" van=""></indien></pre> | |
| Aanvullende informatie is gegeven door: | |
| Naam: | |
| Functie: | |
| Handtekening: | Datum: / / |
| * Doorhalen wat niet van toenassing is | |

De nabestaande krijgt een volledige informatiebrief mee, samen met een kopie van het getekende toestemmingsformulier.

Doorhalen wat niet van toepassing is.